CLINICAL TRIAL: NCT05352672
Title: A Phase 3 Trial of Fianlimab (REGN3767, Anti-LAG-3) + Cemiplimab Versus Pembrolizumab in Patients With Previously Untreated Unresectable Locally Advanced or Metastatic Melanoma
Brief Title: Clinical Study of Fianlimab in Combination With Cemiplimab Versus Pembrolizumab in Adolescent and Adult Patients With Previously Untreated Unresectable Locally Advanced or Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3767-ONC-2011; 2021-004453-23 (EudraCT Number); 2023-505772-30-00 (EU CTIS Number)
Record Dates: First submitted 2022-04-06; First posted 2022-04-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: Unresectable; Metastatic; Stage III; Stage IV; Anti-Lymphocyte-activation gene 3 Pathway (LAG-3)
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — cemiplimab; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A: fianlimab+cemiplimab dose 1 (Experimental): As defined in Protocol Amendment 5
  Interventions: Drug: Fianlimab; Drug: Cemiplimab
- A1: fianlimab+cemiplimab dose 2 (Experimental): As defined in Protocol Amendment 5
  Interventions: Drug: Fianlimab; Drug: Cemiplimab
- B: pembrolizumab+placebo (Experimental): As defined in Protocol Amendment 5
  Interventions: Drug: Pembrolizumab; Drug: Placebo
- C: cemiplimab+placebo (Experimental): As defined in Protocol Amendment 5
  Interventions: Drug: Cemiplimab; Drug: Placebo

INTERVENTIONS:
Drug: Fianlimab — Intravenous (IV) infusion
  Other Names: REGN3767
  Arms: A1: fianlimab+cemiplimab dose 2; A: fianlimab+cemiplimab dose 1
Drug: Cemiplimab — IV infusion
  Other Names: REGN2810; Libtayo
  Arms: A1: fianlimab+cemiplimab dose 2; A: fianlimab+cemiplimab dose 1; C: cemiplimab+placebo
Drug: Pembrolizumab — IV infusion
  Other Names: MK-3475; lambrolizumab; Keytruda
  Arms: B: pembrolizumab+placebo
Drug: Placebo — IV infusion
  Arms: B: pembrolizumab+placebo; C: cemiplimab+placebo

SUMMARY:
This study is researching an experimental drug called REGN3767, also known as fianlimab (R3767), when combined with another medication called REGN2810, also known as cemiplimab (each individually called a "study drug" or called "study drugs" when combined).

The study is focused on patients with a type of skin cancer known as melanoma. The aims of the study are to see how effective the combination of fianlimab and cemiplimab are in treating the melanoma skin cancer, in comparison with a medication, pembrolizumab, approved for the treatment of melanoma skin cancer in adults, and to observe any similarities, or differences, in how the study drugs work in adolescent participants compared with adult participants.

The study is looking at several other research questions, including:

* What side effects may happen from receiving the study drugs
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drugs (which could make the drugs less effective or could lead to side effects). Antibodies are proteins that are naturally found in the blood stream that fight infections.
* How administering the study drugs might improve quality of life

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥12 years on the date of providing informed consent
2. Patients with histologically confirmed unresectable Stage III and Stage IV (metastatic) melanoma (AJCC, 8th revised edition) who have not received prior systemic therapy for advanced unresectable disease

   1. Patients who received adjuvant and/or neoadjuvant systemic therapies are eligible if they did not have evidence of progression or recurrence of disease and/or discontinued due to occurrence of unmanageable imAEs ≥ grade 3 (with the exclusion of endocrinopathies which are fully controlled by hormone replacement) while on such therapies. Also, patients must have had a treatment-free and disease-free interval of >6 months. Accrual of these patients is limited to approximately 10% of the total population enrolled.
   2. Patients with acral and mucosal melanomas are eligible. Accrual will be limited to 10% of the total population.
3. Measurable disease per RECIST v1.1

   1. Previously irradiated lesions can only be counted as target lesions if they have been demonstrated to progress and no other target lesion is available
   2. Cutaneous lesions should be evaluated as non-target lesions
4. Performance status:

   1. For adult patients: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
   2. For pediatric patients: Karnofsky performance status ≥70 (patients ≥16 years) or Lansky performance status ≥70 (patients ≤16 years)
5. Anticipated life expectancy of at least 3 months

Key Exclusion Criteria:

1. Uveal melanoma
2. Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment.
3. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C virus (HCV) infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection
4. Unknown BRAF V600 mutation status as described in the protocol
5. Systemic immune suppression:

   1. Use of immunosuppressive doses of corticosteroids (>10mg of prednisone per day or equivalent) within 14 days of the first dose of study medication. Physiologic replacement doses are allowed up to and including 10mg of prednisone/day or equivalent. Inhaled or topical steroids are permitted, if they are not for treatment of an autoimmune disorder.
   2. Other clinically relevant forms of systemic immune suppression
6. Treatment with other anti-cancer therapy including immuno- therapy, chemotherapy, major surgery or biological therapy within 21 days prior to the first dose of trial treatment. Adjuvant hormonotherapy used for breast cancer or other hormone-sensitive cancers in long term remission is allowed.
7. History or current evidence of significant (CTCAE Grade ≥2) local or systemic infection (e. g., cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 14 days prior to the first dose of trial medication.
8. Active or untreated brain metastases or spinal cord compression. Patients with leptomeningeal disease are excluded. Patients with known brain metastases are eligible if they:

   1. Received radiotherapy or another appropriate standard therapy for the brain metastases,
   2. Have neurologically returned to baseline (except for residual signs and symptoms related to the CNS treatment) for at least 14 days prior to enrollment
   3. Did not require immunosuppressive doses of corticosteroids therapy (>10mg of prednisone per day or equivalent) in the 14 days prior to enrollment
   4. Are asymptomatic with a single untreated brain metastasis <10 mm in size
9. Participants with a history of myocarditis.

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1546 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2031-09-16 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 27 months
  Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on Blinded Independent Central Review (BICR)

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 96 months
Objective response rate (ORR) | Up to 27 months
  Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on Blinded Independent Central Review (BICR) or based on investigator assessment according to RECIST 1.1
Disease control rate (DCR) | Up to 27 months
  Per RECIST 1.1 based on BICR or based on investigator assessment according to RECIST 1.1
Duration of response (DoR) | Up to 27 months
  Per RECIST 1.1 via BICR or based on investigator assessment according to RECIST 1.1
PFS | Up to 27 months
  Based on investigator assessment according to RECIST 1.1
Incidence of Adverse Events (AEs) | Up to 90 days post last dose, approximately 6 years
  Including treatment emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), and/ or immune-mediated adverse events (imAEs)
Occurrence of interruption and discontinuation of study drug(s) due to AEs | Up to 90 days post last dose, approximately 6 years
  Including TEAEs, AESIs, and/ or imAEs
TEAEs leading to death | Up to 6 years
Incidence of laboratory abnormalities | Up to 90 days post last dose, approximately 6 years
  Will be graded using the current version of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grading system (version 5.0)
Concentrations of cemiplimab in serum | Up to 90 days post last dose, approximately 6 years
Concentrations of fianlimab in serum | Up to 90 days post last dose, approximately 6 years
Incidence of anti-drug antibodies (ADA) to fianlimab over time | Up to 30 days post last dose, approximately 6 years
Titer of anti-drug antibodies (ADA) to fianlimab over time | Up to 30 days post last dose, approximately 6 years
Incidence of ADA to cemiplimab over time | Up to 30 days post last dose, approximately 6 years
Titer of ADA to cemiplimab over time | Up to 30 days post last dose, approximately 6 years
Incidence of neutralizing antibodies (NAb) to fianlimab over time | Up to 30 days post last dose, approximately 6 years
Incidence of NAb to cemiplimab over time | Up to 30 days post last dose, approximately 6 years
Patient-reported outcomes (PROs) as measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) | Up to 90 days post last dose, approximately 6 years
  EORTC-QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
PROs as measured by EQ-5D-5L | Up to 90 days post last dose, approximately 6 years
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Overall scores range from 0 to 1, with low scores representing a higher level of dysfunction.
PROs as measured by Functional Assessment of Cancer Therapy melanoma (FACTM) (melanoma subscale only) | Up to 90 days post last dose, approximately 6 years
  The FACTM is a melanoma-specific quality of life questionnaire that is composed of items from the Functional Assessment of Cancer Therapy-General (FACT-G). The FACTM is scored on a 5 point Likert-scale: "Not at all", "A little bit", "Somewhat", "Quite a bit", and "Very much.". A Higher score represents higher Health Related Quality of Life (HRQoL).
PROs as measured by Patient Global Impression of Severity (PGIS) | Up to 21 days post last dose, approximately 6 years
  The PGIS is a single 1-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time by using a 4-point Likert scale that ranges from (1) = "none (no symptoms)" to (4) = "severe".
PROs as measured by Patient Global Impression of Change (PGIC) | Up to 21 days post last dose, approximately 6 years
  The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change since starting treatment as rated on a 5-point Likert scale anchored by (1) "much better" to (5) "much worse", with (4) = "no change"
Change in physical functioning per EORTC QLQ-C30 | Baseline to Week 25
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in role functioning per EORTC QLQ-C30 | Baseline to Week 25
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in global health status/quality of life (GHS/QoL) per EORTC QLQ-C30 | Baseline to Week 25
  Global Health Status/Quality of Life (GHS/Qol) Score (Items 29 and 30) using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in physical functioning per EORTC QLQ-C30 | Baseline to end of study, approximately 6 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in role functioning per EORTC QLQ-C30 | Baseline to end of study, approximately 6 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in GHS/QoL per EORTC QLQ-C30 | Baseline to end of study, approximately 6 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (210):
- United States (5):
  - UC San Diego, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Orlando Health, Orlando, Florida
  - Seidman Cancer Center, Cleveland, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
- Argentina (6):
  - DIABAID - Instituto de Asistencia Integral en Diabetes, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Medico Austral, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro de Investigacion Pergamino, Pergamino, Buenos Aires
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas y Desarrollo LC S.R.L. (LC Investigacion), Buenos Aires
  - Exelsus, San Miguel de Tucumán
- Australia (6):
  - Gold Coast Hospital and Health Service, Southport, Queensland
  - Townsville University Hospital, Townsville, Queensland
  - Calvary North Adelaide Hospital, North Adelaide, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Andrew Love Cancer Centre, Geelong, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Austria (4):
  - University Hospital Saint Poelten, Sankt Pölten, Lower Austria
  - Medical University of Graz, Graz, Styria
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Medical University Vienna, Vienna
- Belgium (4):
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - AZ Nikolaas, Sint-Niklaas, West-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire Universite Catholique de Louvain Namur Site Sainte Elisabeth, Namur
- Brazil (20):
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Hospital das Clinicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Liga Paranaense de Combate ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Instituto do Cancer em Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de vento, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Amor Amazonia, Porto Velho, Rondônia
  - Catarina Pesquisa Clinica, Itajaí, Santa Catarina
  - Instituto Joinvilense de Hematologia e Oncologia, Joinville, Santa Catarina
  - Animi Unidade de Tratamento Oncologico, Lages, Santa Catarina
  - Fundacao Pio XII - Hospital de Amor, Barretos, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Oncosite Centro De Pesquisa Em Oncologia, Ijuí
  - INCA - Brazilian National Cancer Institute, Rio de Janeiro
  - Instituto COI, Rio de Janeiro
  - Hemomed, São Paulo
  - Hospital Sirio Libanes, São Paulo
  - Sao Camilo Oncologia, São Paulo
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Dr. Everett Chalmers Hospital, Fredericton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Chile (6):
  - Hospital Clinico Universidad de Chile, Santiago, Independencia
  - Oncocentro APYS, Viña del Mar, Región de Valparaíso
  - Centro Oncologia de Precision Universidad Mayor, Santiago, Santiago Metropolitan
  - Oncovida, Santiago, Santiago Metropolitan
  - Centro Oncologico del Norte, Antofagasta
  - Bradford Hill, Santiago
- Czechia (3):
  - University Hospital Hradec Kralove, Hradec Králové, North Central Czech Republic
  - Fn Kralovske Vinohrady, Dermatological Clinic, Vinohrady, Prague
  - University Hospital Ostrava, Ostrava
- France (19):
  - Hospices Civils de Lyon, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU-Dijon, Dijon, Burgundy
  - Besancon Regional University Hospital Center, Besançon, Doubs
  - Chu De Bordeaux, Bordeaux, Gironde
  - Centre Hospitalier Universitaire (CHU) de Lille, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche, Isere
  - CHU Charles Nicolle, Rouen, Normandy
  - Centre Hospitalier Universitaire De Poitiers, Poitiers, Nouvelle-Aquitaine
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - CHU de St Etienne, Saint Priest En Jarez, Pays de la Loire Region
  - Gustave Rroussy, Villejuif, Val de Marne / Ile de France
  - Hopital Ambroise Pare, Boulogne
  - CHU Estaing, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Nantes University Hospital, Nantes
  - Clinique Sainte Anne, Strasbourg
  - Hopital Avicenne, Bobigny, Île-de-France Region
  - Hospital Henri Mondor, Créteil, Île-de-France Region
  - Cochin Hospital, Paris, Île-de-France Region
- Georgia (8):
  - Cancer Center of Adjara, Batumi
  - Acad.Fridon Todua Medical Center- Research Institute of Clinical Medicine, Tbilisi
  - Israeli Georgian Medical Research Clinic Helsicore, Tbilisi
  - LTD New Hospitals, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - TIM - Tbilisi Institute of Medicine, Tbilisi
  - ltd Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (21):
  - University Medical Center Mannheim, Mannheim, Baden-Wurttemberg
  - University of Tuebingen, Tübingen, Baden-Wurttemberg
  - LMU Klinikum, Munich, Bavaria
  - Klinikum Nurnberg, Hautklinik, Universitatsklinik fur Dermatologie der Paracelsus Medizinischen Privatuniversitat, Nuremberg, Bavaria
  - University Hospital of Regensburg, Regensburg, Bavaria
  - University Clinic Frankfurt, Frankfurt am Main, Hesse
  - University Hospital Giessen, Giessen, Hesse
  - Elbekliniken Stade Buxtehude, Buxtehude, Lower Saxony
  - Ruhr University Bochum, Bochum, North Rhine-Westphalia
  - Fachklinik Hornheide, Münster, North Rhine-Westphalia
  - Universitatsmedizin der Johannes-Gutenberg Universitat Mainz, Mainz, Rhineland-Palatinate
  - University Hospital Dresden, Dresden, Saxony
  - Universitatsklinikum Leipzig, AoR, Leipzig, Saxony
  - Dermatologie, Dessau, Saxony-Anhalt
  - Skin Cancer Center Harz, Quedlinburg, Saxony-Anhalt
  - University Hospital of Universitatsklinikum Schleswig Holstein (UKSH) Campus Kiel, Kiel, Schleswig-Holstein
  - Universitatsklinikum Schleswig Holstein Campus Luebeck, Lübeck, Schleswig-Holstein
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - Charite Universitaetsmedizin Berlin, Berlin
  - University Medical Center Gottingen, Göttingen
  - Helios Kliniken Schwerin, Schwerin
- Hungary (3):
  - University of Pecs Medical School, Pécs, Baranya
  - University of Debrecen, Debrecen, Hajdú-Bihar
  - Szabolcs Szatmar Bereg Megyei Korhazak Es Egyetemi Oktatokorhaz, Nyíregyháza, Szabolcs-Szatmár-Bereg
- Ireland (4):
  - Galway University Hospital, Galway, Connacht
  - Cork University Hospital, Cork
  - Tallaght University Hospital, Dublin
  - St Vincents University Hospital, Dublin
- Italy (21):
  - U.O.C. Oncologia Medica ed Ematologia (U.O.C Medical Oncology and Hematology), Naples, Campania
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Istituto Clinico Humanitas, Rozzano, Milan
  - FPO IRCCS Candiolo, Candiolo, Torino
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Istituto dei Tumori, Bari
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Santa Croce i Carle, Cuneo
  - Fondazione IRCCS Istituto Nazionale dei Tumori., Milan
  - Istituto Europeo di Oncologia, Milan
  - Universita Degli Studi Di Milano-Bicocca - Azienda Ospedaliera San Gerardo Di Monza, Monza
  - Istituto Nazionale Tumori IRCCS Fondazione G Pascale, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carita - Oncology, Novara
  - Vento Institute of Oncology IOV-IRCCS, Padua
  - Campus Bio-Medico di Roma, Rome
  - IRCCS Regina Elena National Cancer Institute, Rome
  - Istituto Dermopatico dell'Immacolata, Rome
  - Aou Citta della Salute e della Scienza di Torino - SC Dermatologia U, Torino
  - Santa Chiara Hospital, Trento
  - Azienda Sanitaria Universitaria del Friuli Centrale, Udine
- Mexico (9):
  - Centro De Estudios Y Prevention Del Cancer, Tuxtla Gutiérrez, Chiapas
  - Preparaciones Oncologica SC, León, Guanajuato
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos SA de CV, Zapopan, Jalisco
  - iCan Oncology, Monterrey, Nuevo León
  - Neurociencias Estudios Clinicos SC, Culiacán, Sinaloa
  - Centro De Atencion E Investigacion Clinica En Oncologia SCP, Mérida, Yucatán
  - Centro Estatal de Cancerologia, Chihuahua City
  - FAICIC S. de R.L. de C.V., Veracruz
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Centre Groningen, Groningen
- Peru (8):
  - Instituto Regional de Enfermedades Neoplasicas del Centro - IREN CENTRO, Concepción, Departamento de Junín
  - Clinica Peruano Americana (Private practice), Trujillo, La Libertad
  - Clinica Oncosalud, San Borja, Lima region
  - Instituto Nacional de Enfermedades Neoplasicas, Surquillo, Lima region
  - Hospital Nacional Daniel A. Carrion, Lima, Provincia Constitucional del Callao
  - Hospital Goyeneche, Arequipa
  - Centro Medico Monte Carmelo, Arequipa
  - Clinica Internacional SA, Lima
- Poland (5):
  - Mazowiecki Szpital Wojewodzki, Siedleckie Centrum Onkologii, Siedlce, Mazxowieckie
  - Uniwersyteckie Centrum Kliniczne (UCK), Gdansk, Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Słupsk, Pomeranian
  - Poznan University of Meidcla Science, Poznan, Wielkopolska
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Romania (10):
  - Institute of Oncology Bucharest, Bucharest, București
  - Cardiomed, Cluj-Napoca, Cluj
  - Medisprof, Cluj-Napoca, Cluj
  - Radiotherapy Center Cluj, Floreşti, Cluj
  - Sfantul Nectarie Oncology Center, Craiova, Dolj
  - SC RTC Radiology Therapeutic Center SRL, Otopeni, Ilfov
  - Oncocenter Oncologie Clinica S.R.L, Timișoara, Timiș County
  - Oncomed, Timișoara, Timiș County
  - Centrul De Oncologie Euroclinic, Iași
  - Regional Institute of Oncology, Iași
- South Africa (3):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Cape Town Oncology Trials, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
- Spain (21):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - H. Germans Trias i Pujol, ICO-Badalona, Badalona, Barcelona
  - Instituto Oncologico Dr Rosell Hospital Universitari Quiron Dexeus Location, Barcelona, Catalonia
  - Onkologikoa, Donostia / San Sebastian, Gipuzkoa
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Teresa Herrera-Chuac, A Coruña, Spain/La Coruna
  - Catalan Institute of Oncology (ICO) Hospitalet, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Catalan Institute Of Oncology, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Pa<, Madrid
  - Centro Integral Oncologico HM Clara Campal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - Incliva - Instituto de Investigacion Sanitaria, Valencia
- Turkey (Türkiye) (13):
  - Baskent University, Yüreğir, Adana
  - Medical oncology, Istanbul, Bakirkoy
  - Ege University, Izmir, Bornova
  - Kocaeli University, İzmit, Kocaeli
  - Gaziantep Medicalpoint Hospital, Gaziantep, Sehitkamil
  - Gulhane Training and Research Hospital, Ankara
  - Ozel Liv Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Dicle University - Medical Faculty Campus, Diyarbakır
  - Trakya University, Edirne
  - Bezmialem University, Istanbul
  - Istanbul University Cerrahpasa at Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Medeniyet University - Prof Dr Suleyman Yalcin Sehir Hospital, Istanbul
- United Kingdom (4):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Hull University Teaching Hospitals NHS Trust, Cottingham, East Yorkshire
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - Royal Surrey County Hospital, Guildford

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: A clinical study for adults and adolescents with advanced melanoma skin cancer. — https://harmonymelanomastudy.com/